CLINICAL TRIAL: NCT02220439
Title: Nested Case-control Analysis of the Influence of the Microbiome on Rotavirus Vaccine Immunogenic Response in Infants in Karachi, Pakistan
Brief Title: Does the Fecal Microbiome Influence Rotarix Immunogenicity
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Aga Khan University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); University of Padova (Other); Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Vanessa Harris, V.C. Harris, M.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AIGHD-CSP2013-001a
Record Dates: First submitted 2014-06-10; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Rotavirus Infections; Reaction - Vaccine Nos; Intestinal Bacteria Flora Disturbance
Keywords: rotavirus; immunogenicity; enteric vaccine; vaccine immunogenicity; rotavirus vaccine; gut microbiome; microbiome
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: non-rotavirus seroconverters: Infants not demonstrating seroconversion to rotavirus vaccination, as measured anti-RV Immunoglobulin A < 20 U/ml
- Control: rotavirus seroconverters: Infants demonstrating seroconversion to rotavirus vaccination, as measured by anti-rotavirus Immunoglobulin A > 20 U/ml

SUMMARY:
This is a proposal for a nested case-control study within an ongoing rotavirus vaccine immunogenicity clinical trial Karachi, Pakistan. The primary study aim is to compare the fecal microbiota composition and diversity of infants who do (control) and do not (case) demonstrate immune seroconversion to rotavirus vaccination. The infants will be matched for vaccination dose, age and breast-feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks 0 days to 7 weeks 6 days age at the time of enrollment.
* Healthy infant free of chronic or serious medical condition as determined by history and physical exam at time of enrollment into in the study.
* Written informed consent obtained from the parents or guardians.
* Availability of baseline fecal sample collected before Rotarix vaccination
* Written informed consent obtained from the parents or guardians for nested study

Exclusion Criteria:

* Hypersensitivity to any of the vaccine components
* Use of any investigational drug or vaccine other than the study vaccine within 30 days of first dose of study vaccine or during the study.
* Use of any immunosuppressive drugs.
* Previous intussusceptions or abdominal surgery.
* Enrollment in any other trial (besides NCT01199874).
* Birth weight less than 1500 grams; or if birth weight is unknown, weight less than 2000 grams on or before 28 days.
* Immunoglobulin and/or blood products use since birth or during the study period. Nested study additional exclusion criteria:
* Positive serum anti-rotavirus Immunoglobulin A (> 20 U/ml) at 6 weeks of age, indicative of prior rotavirus infection

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be nested within an existing rotavirus immunogenicity study being conducted in Karachi, Pakistan (clinicaltrials.gov: NCT01199874) . The physical setting is a peri-urban slum outside of Karachi, primarily populated by fishermen. Parents and legal guardians of infants participating in NCT01199874 will provide new informed consent for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
microbiome diversity (Shannon's index) and composition (relative abundance) | at 6 weeks of age, pre-rotavirus vaccination
  Microbiota composition will be measured by calculating and comparing a % of the phylogenetic groups present in both groups
  Diversity will be measured by calculating a comparing a Shannon's reciprocal index of diversity, 1/D in both groups
  The relative abundance of microbial groups will be measured by calculating and comparing the ribosomal ribonucleic acid gene copy per gram of feces over time in both groups

SECONDARY OUTCOMES:
microbiome diversity (Shannon's index) and composition (relative abundance) | at 1 to 3 years of age post-rotavirus vaccination
  Microbiota composition post vaccination will be measured by calculating and comparing a % of the phylogenetic groups present in both groups
  Diversity post vaccination will be measured by calculating a comparing a Shannon's reciprocal index of diversity, 1/D in both groups
  The relative abundance of microbial groups post vaccination will be measured by calculating and comparing the ribosomal ribonucleic acid gene copy per gram of feces over time in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa C Harris, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)